CLINICAL TRIAL: NCT00244790
Title: The Effects of Obesity and Protein Intake on the Kidney
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Allon Friedman, MD, MD, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0309-03; K23RR019615-01A1 (NIH)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Diseases
Keywords: glomerular hyperfiltration; proteinuria
MeSH Terms: conditions — Kidney Diseases; Proteinuria | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- low protein (Experimental)
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — crossover low vs high protein diet before and after weight loss
  Other Names: Diet 1; Diet 2

SUMMARY:
The purpose of this study is to determine if being overweight and eating lots of protein causes separate changes in the kidney that lead to kidney disease over time. These questions are important because the number of people who have kidney disease is quickly growing. If being overweight and eating lots of protein is found to cause kidney disease, then doctors may be able to limit the number of people with kidney disease by recommending weight loss and eating less protein

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that being obese leads to changes in kidney function that are independent of, and enhanced by, high dietary protein intake. Kidney function will be measured by the kidney's ability to filter blood and by the amount of protein in the urine. The hypothesis will be tested in the following manner: The first part of the study will involve a crossover design comparing kidney function in obese people with stable weights on a low and high protein diet ("Low/High Protein Study"). The second part of the study will compare kidney function in obese people before and after weight reduction surgery ("Before/After Surgery Study"). Since certain changes in kidney function may lead to kidney disease over time, it is important to confirm the effects of obesity and dietary protein intake on the kidney, especially with the current rise in obese people and the popularity of high protein diets.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Ability to give informed consent
* Not pregnant and using appropriate contraceptive methods, or not of childbearing potential
* BMI of 30 or higher

Exclusion Criteria:

* Iodine or shellfish allergy
* History of adverse reaction to intravenous contrast
* Dialysis dependence
* Diagnosis of diabetes mellitus or taking medicine for diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
glomerular filtration rate | days

CONTACTS AND LOCATIONS:
Overall Officials: Allon Friedman, MD, Principal Investigator — Indiana University
Locations (1):
- University Hospital, Indianapolis, Indiana, United States